CLINICAL TRIAL: NCT00778570
Title: A Combined Retrospective and Prospective Chart Review Analysis of Visual Outcomes Following Excimer Laser Vision Correction
Brief Title: Advanced Surface Ablation (ASA) vs Laser-Assisted In Situ Keratomileusis (LASIK)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2006800-01H
Record Dates: First submitted 2008-10-21; First posted 2008-10-23 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Nearsightedness; Farsightedness; Astigmatism
MeSH Terms: conditions — Myopia; Hyperopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ASA: Participants treated for Excimer laser vision correction using Advanced Surface Ablation (ASA).
- LASIK: Participants treated for Excimer laser vision correction using Laser-Assisted In Situ Keratomileusis (LASIK)

SUMMARY:
The purpose of this combined retrospective and prospective chart review analysis is to investigate the safety, efficacy, and predictability obtained via Laser-Assisted In Situ Keratomileusis (LASIK) and Advanced Surface Ablation (ASA) over a wide range of refractive errors

The working hypothesis is that there will be no difference in clinical outcomes between patients treated with LASIK or ASA.

DETAILED DESCRIPTION:
Excimer laser vision correction (LVC) is a widely used procedure to correct nearsightedness, farsightedness, and astigmatism by reshaping the surface of the eye (cornea). Laser-Assisted In Situ Keratomileusis (LASIK) and Advanced Surface Ablation (ASA) and are techniques currently used to prepare the cornea for Excimer LVC.

This review is intended to study whether LASIK is equal in visual outcome (null hypothesis), more effective (alternate hypothesis 1) or less effective (alternate hypothesis 2) than ASA in clinical outcome up to one year.

ELIGIBILITY:
Inclusion Criteria:

* Eyes that were treated for LASIK or ASA Excimer laser vision correction before December 1st 2006 and newly recruited eyes that qualify for LASIK or ASA Excimer laser vision correction may be enrolled in this study.

Exclusion Criteria:

* There are no exclusion criteria; all patients that went forward with Excimer laser vision correction may be included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female participants from the Ottawa/Gatineau region requesting laser vision correction to correct nearsightedness, farsightedness, and/or astigmatism.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2007-02; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | 1 day, 1W, 1M, 3M, 6M, 9M, 12M

CONTACTS AND LOCATIONS:
Overall Officials: George Mintsioulis, MD, Principal Investigator — University of Ottawa Eye Institute
Locations (1):
- University of Ottawa Eye Institute, Ottawa, Ontario, Canada